CLINICAL TRIAL: NCT03106155
Title: Phase II, Single-arm Study of Vistusertib (AZD2014) Monotherapy in Relapsed Small Cell Lung Cancer Patients Harboring RICTOR Amplification(SUKSE-D)
Brief Title: Vistusertib (AZD2014) Monotherapy in Relapsed Small Cell Lung Cancer Patients Harboring RICTOR Amplification
Acronym: [SUKSES-D]
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of IP support organization
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Keunchil Park, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01-003
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — vistusertib

STUDY DESIGN:
Intervention Model Description: Vistusertib monotherapy (50 mg BID per os every 12 hours)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vistusertib (AZD2014) (Experimental): vistusertib (AZD2014), 50 mg,BID, per os, every 12 hours
  Interventions: Drug: vistusertib (AZD2014)

INTERVENTIONS:
Drug: vistusertib (AZD2014) — vistusertib(AZD2014): 50 mg BID per os every 12 hours administration daily. One cycle is consisted of 3 weeks.

SUMMARY:
[Study Design] This study is a single arm, multi-center phase II study of vistusertib monotherapy in patients with relapsed small cell lung cancer (SCLC) harboring RICTOR amplification. Patients will receive vistusertib monotherapy (50 mg BID per os every 12 hours) until they demonstrate objective disease progression or they meet any other discontinuation criteria.

[Primary Objective] To investigate the efficacy of vistusertib monotherapy in patients with relapsed SCLC patients harboring RICTOR amplification as 2nd or 3rd line therapy

ELIGIBILITY:
[Inclusion Criteria]

* Provision of informed consent prior to any study specific procedures
* Men and women aged at least 18 years
* Small cell lung cancer harboring RICTOR amplification
* Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with no deterioration over the previous 2 weeks
* Minimum life expectancy of 12 weeks
* Patients must have acceptable bone marrow, liver and renal function measured within 14 days prior to administration of study treatment as defined below:
* At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and follow up visits.
* No history of non-autologous bone marrow transplant.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 21 days.
* Prior chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents within 21 days of starting study treatment. Prior use of an investigational monoclonal antibody therapy within 3 months.
* Major surgery within 4 weeks prior to study entry (excluding placement of vascular access), or minor surgery (excluding tumour biopsies) within 14 days of first dose of study treatment.
* Exposure to strong or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP if taken within the stated washout periods before the first dose of study treatment (see Appendix 1)
* Exposure to specific substrates of the drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K within the appropriate wash-out period
* Any haemopoietic growth factors within 14 days prior to receiving study treatment.
* Pre-treatment with other PI3K, AKT, dual PI3K/mTRO and mTOR inhibitors
* Spinal cord compression and/or brain metastases unless asymptomatic or treated and stable off steroids for at least 4 weeks prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) by RECIST 1.1 | Up to 20 months
  Assessments to be performed using CT or MRI scans. To be measured according to RECIST 1.1

SECONDARY OUTCOMES:
Duration of response | Up to 20 months
  Assessments to be performed using CT or MRI scans. To be measured according to RECIST 1.1
Disease control rate | at 12 weeks
  Assessments to be performed using CT or MRI scans. To be measured according to RECIST 1.1
Overall survival (OS) | Up to 20 months
  Kaplan-Meier method
Progression-free survival (PFS) | Up to 20 months
  Kaplan-Meier method
Number of participants with Adverse Events as Assessed by CTCAE v4.03 | Up to 20 months
  CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical center, Seoul, South Korea